CLINICAL TRIAL: NCT06412640
Title: Eradication of Helicobacter Pylori by 14-day Dual Therapy of Keverprazan in Combination With Low-dose and High-dose Amoxicillin: a Prospective, Single-center, Developmental-label, Randomized Controlled Study
Brief Title: Optimization of Keverprazan-amoxicilli Dual Therapy for Helicobacter Pylori
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20240419-15
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: H. Pylori Infection
MeSH Terms: interventions — Amoxicillin; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high dose amoxicillin with keverprazan group (Active Comparator): Patients need to take keverprazan 20mg bid and amoxicillin 1000mg tid for 14 days.
  Interventions: Drug: Keverprazan; Drug: Amoxicillin
- low dose amoxicillin with keverprazan group (Experimental): Patients need to take keverprazan 20mg bid and amoxicillin 1000mg bid for 14 days.
  Interventions: Drug: Keverprazan; Drug: Amoxicillin

INTERVENTIONS:
Drug: Keverprazan — Potassium-competitive acid blocker
  Other Names: Potassium-competitive acid blocker
Drug: Amoxicillin — Antibiotic for H. pylori eradication
  Other Names: Antibiotic for H. pylori eradication

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of keverprazan with different doses of amoxicillin for Helicobacter Pylori.

DETAILED DESCRIPTION:
This study is a prospective, single-center, open-label, randomized, parallel-controlled trial. A total of 268 H. pylori positive patients needed to be recruited and were randomized into 2 groups in 1:1 ratio, Group A was the control group and subjects were required to take keverprazan 20mg,bid and amoxicillin 1.0g,tid for 14 days. Group B was the experimental group and subjects were required to take keverprazan 20mg,bid and amoxicillin 1.0g,tid for 14 days. All the above regimens were used for eradication of H. pylori. During the 14-day eradication treatment, all subjects were instructed and asked to record their adverse drug reactions and compliance. On days 7 and 14 of treatment, researchers followed up with patients via WeChat or phone to determine adverse reactions and compliance, and observed and recorded whether subjects experienced any adverse reactions such as nausea, diarrhea, dizziness, bitter taste in the mouth, rash, and constipation. Subjects were seen again 4 weeks after the end of treatment to check for H. pylori eradication by 13C-UBT or 14C-UBT. Patients were encouraged, but not required, to undergo tongue and fecal flora testing before and after H. pylori eradication to determine the short-term effects of different doses of amoxicillin in combination with keverprazan for 14 days on the patient's tongue and intestinal flora.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Helicobacter pylori positivity through 13C-UBT or 14C-UBT
2. Patients who have not received eradication treatment for Helicobacter pylori in the past, or who have failed eradication in the early stage but have not received eradication treatment within six months
3. Voluntarily participate in this experiment and sign an informed consent form

Exclusion Criteria:

1. Allergies to research drugs (such as those allergic to penicillin, amoxicillin, keverprazan)
2. Patients with peptic ulcer
3. Patients who have received Helicobacter pylori eradication treatment within six months
4. Use antibiotics or bismuth medication 4 weeks before starting the study；use P-CAB or PPI 2 weeks before starting the study
5. Using corticosteroids, non steroidal anti-inflammatory drugs, or anticoagulants
6. Those who are using atazanavir, nelfinavir, rilpivirine, itraconazole, tyrosine kinase inhibitors (imatinib, gefitinib, etc.), digoxin, and methyl digoxin
7. History of esophageal or gastric surgery
8. Pregnant or lactating women
9. Suffering from serious concomitant diseases such as liver disease, cardiovascular disease, lung disease, or kidney disease
10. Excessive drinking
11. Gastric mucosa-associated lymphoid tissue lymphoma (MALT), malignant neoplastic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | at least four weeks after completion of the medication
  Subjects were seen again 4 weeks after the end of treatment to check for H. pylori eradication by 13C-UBT or 14C-UBT.

SECONDARY OUTCOMES:
Adverse even | Within 7 days after completion of therapy
  Adverse drug reactions are classified into six types: dose-related, non-dose-related, dose-related and time-related, time-related, withdrawal, and failure of therapy.
Compliance Rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, Principal Investigator — Nanjing First Hospital, Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Choi H, Leung K, Jiang F, Graham DY, Leung WK. Global prevalence of Helicobacter pylori infection between 1980 and 2022: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2023 Jun;8(6):553-564. doi: 10.1016/S2468-1253(23)00070-5. Epub 2023 Apr 20. PMID 37086739
- [Background] Zhou XZ, Lyu NH, Zhu HY, Cai QC, Kong XY, Xie P, Zhou LY, Ding SZ, Li ZS, Du YQ; National Clinical Research Center for Digestive Diseases (Shanghai), Gastrointestinal Early Cancer Prevention & Treatment Alliance of China (GECA), Helicobacter pylori Study Group of Chinese Society of Gastroenterology and Chinese Alliance for Helicobacter pylori Study.. Large-scale, national, family-based epidemiological study on Helicobacter pylori infection in China: the time to change practice for related disease prevention. Gut. 2023 May;72(5):855-869. doi: 10.1136/gutjnl-2022-328965. Epub 2023 Jan 23. PMID 36690433
- [Background] Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Online ahead of print. PMID 35944925
- [Background] Hu Y, Xu X, Ouyang YB, He C, Li NS, Xie C, Peng C, Zhu ZH, Xie Y, Shu X, Lu NH, Zhu Y. Optimization of vonoprazan-amoxicillin dual therapy for eradicating Helicobacter pyloriinfection in China: A prospective, randomized clinical pilot study. Helicobacter. 2022 Aug;27(4):e12896. doi: 10.1111/hel.12896. Epub 2022 Apr 25. PMID 35466521
- [Background] Zhou S, Xie L, Zhou C, Wang L, Chen J, Ding S, Zhu B, Su M, Shao F. Keverprazan, a novel potassium-competitive acid blocker: Multiple oral doses safety, tolerability, pharmacokinetics, and pharmacodynamics in healthy subjects. Clin Transl Sci. 2023 Oct;16(10):1911-1922. doi: 10.1111/cts.13598. Epub 2023 Aug 2. PMID 37533172